CLINICAL TRIAL: NCT04528758
Title: Preliminary Evaluation of F-18 Rhodamine 6G in Healthy Individuals and Patients With Stable Heart Condition
Brief Title: F-18 Rhodamine 6G PET Imaging for Myocardial Blood Flow
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: re-evaluation of radiotracer
Sponsor: Washington University School of Medicine (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201808025
Record Dates: First submitted 2020-08-13; First posted 2020-08-27 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — rhodamine 6G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dosimetry group (Experimental): Patients in the dosimetry group will be imaged with the radio-pharmaceutical Rhodamine 6G at different time points. 0-120, 30-150, 60-180
  Interventions: Drug: Rhodamine 6G
- Stable Heart Patients (Active Comparator): Stable heart patients will be given a rest/stress PET/CT with Rhodamine 6G myocardial perfusion study to determine myocardial blood flow
  Interventions: Drug: Rhodamine 6G

INTERVENTIONS:
Drug: Rhodamine 6G — Rhodamine 6G radio-pharmaceutical will be injected to determine myocardial blood flow
  Other Names: PET/positron Emission Tomography imaging

SUMMARY:
Use of novel radio-pharmaceutical Rhodamine 6G to determine myocardial blood flow

DETAILED DESCRIPTION:
Using Rhodamine 6G to determine myocardial blood flow in normal volunteers and patients with coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 21-75 years of age and any race.
* Capable of giving written informed consent.
* "Healthy adult volunteer subject" is someone who is volunteering to undergo imaging procedures and based on screening procedures has no known significant health problems.
* Stable patients with known or suspected coronary artery disease that are scheduled to have or have undergone a clinically indicated conventional rest/stress SPECT MPI and no intervention between SPECT and PET.
* Female subjects must not be pregnant or lactating.

Exclusion Criteria:

* Has any condition that, in the opinion of the Sponsor-Investigator or designee could increase risk to the subject, limit the subject's ability to tolerate the research procedures, or interfere with collection of the data.
* Have abnormal findings on any screening/baseline procedure, e.g. physical examination, laboratory tests, electrocardiogram that suggest the subject might have a condition that could, in the opinion of the Sponsor-Investigator, affect the subject's response to the radiopharmaceutical or related research procedures.
* Is deemed likely to be unable to perform all research procedures for any reason, (e.g., subjects unable to lie still or inability to tolerate up to 60 minutes in a supine position with arms up during the PET imaging procedures due to chronic back/shoulder pain or arthritis as assessed by physical examination and medical history).
* Has a history of hypersensitivity to Fluorine-18 or other radiopharmaceutical or any of its excipients.
* Have contraindications to cardiovascular PET/CT imaging such as claustrophobia.
* Have high blood pressure (>200/110)
* Have Epilepsy
* Have major kidney or liver problems
* Have current or past history of major medical illness
* Currently using recreational drugs
* Body weight of > 300 lbs. (weight limit of the PET/CT table)
* Stable Cardiac Disease: Rest/Stress Group only:

  * Cardiac patients who suffer an intervening clinical event such as worsening angina pectoris or myocardial infarction or whom undergo a myocardial revascularization procedure or have myocardial ischemia at rest.
  * Sinus node disease (e.g. SA block) or symptomatic bradycardia, second or third degree atrioventricular (AV) block.
  * Pre-existing obstructive lung disease (e.g. asthma) that precludes the safe administration of the pharmacological stressor according to the approved label.
  * Uncontrolled and severe hypertension (e.g. systolic blood pressure >200 mmHg, diastolic blood pressure >110 mmHg).
  * Baseline hypotension (e.g. systolic blood pressure < 90 mmHg, diastolic blood pressure <50 mmHg).
  * Seizures
  * The use of caffeine, nicotine or over the counter cold medicines within 12 hours prior to stress imaging day with regadenoson.
  * The theophylline-based medications or dipyridamole within 48 hours prior to each imaging day.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dosimetry group | 1-2 days
  Evaluate both image quality and myocardial blood flow at different imaging time points.
  Image quality provides higher count Density and high spatial resolution, which makes it easier to see the heart vessels, and myocardial blood flow is measured in mL/g/min. Both measurements will be agregated to arrive at one reported value helps determine the balance of heart disease and in small and large vessels

SECONDARY OUTCOMES:
Stable Heart Patients | 1-2 days
  Determine myocardial blood flow in stable heart patients. Myocardial blood flow is measured in mL/g/min which can show normal blood flow with stable patients.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gropler, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided